CLINICAL TRIAL: NCT01534689
Title: An Evaluation of the Effect of the Erchonia FX-405™ on Treating Toenail Onychomycosis Clinical Study
Brief Title: Study of the Use of Low Level Laser Light Therapy to Treat Toenail Fungus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC_TF_001
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erchonia FX-405™ Laser (Experimental): The Erchonia FX-405™ Laser is a dual-diode laser emitting 15.5-17.5 milliWatts (mW) of 635 nanometer (nm) red laser light and 23.5-25.5 mW 405 nm blue laser light. The the power reaching the surface of the skin is 1 mW
  Interventions: Device: Erchonia FX-405™ Laser

INTERVENTIONS:
Device: Erchonia FX-405™ Laser — The Erchonia FX-405™ dual diode laser light is directed at the great toenail at a distance of approximately 6 inches above the toenail. The dual wavelengths of 405 nm and 635 nm are activated simultaneously for 10 minutes of total treatment administration time.

SUMMARY:
The purpose of this study is to determine whether low level laser light is effective in the treatment of toenail fungus.

DETAILED DESCRIPTION:
An infection of toenail fungus, or onychomycosis, occurs when fungi infect one or more nails. As the nail fungus spreads deeper into the nail, it may cause nail discoloration, thickening and the development of crumbling edges, all of which can lead to an unsightly and potentially painful problem. Onychomycosis is difficult to treat, and infections recur easily. Toenail fungus affects approximately 23 million people in the US - about 10% of all adults. Currently available treatments for toenail fungus are lacking. Even the most effective oral medications are successful only about half of the time. Topical medications are successful less than 10% of the time. Recently, research has found laser therapy to show promise as a novel alternative treatment for toenail onychomycosis. Unlike medication-driven treatments for toenail fungus which can have many side effects including serious ones such as liver toxicity, laser therapy presents minimal risk of side effects. Laser therapy is applied to toenail onychomycosis by shining a laser light through the toenail. The laser light vaporizes the fungus while leaving the skin and surrounding tissue unharmed.

ELIGIBILITY:
Inclusion Criteria:

* Onychomycosis present in at least one great toenail.
* Disease involvement is at least 25%.
* Subject is willing and able to refrain from employing other (non-study) treatments (traditional or alternative) for his or her toenail onychomycosis throughout study participation.
* Subject is willing and able to refrain from the use of nail cosmetics such as clear and/or colored nail lacquers throughout study participation.

Exclusion Criteria:

* Spikes of disease extending to nail matrix.
* Infection involving lunula, e.g., genetic nail disorders, primentary disorders.
* Less than 2mm clear (unaffected) nail plate length beyond the proximal fold.
* Presence of dermatophytoma (thick masses of fungal hyphae and necrotic keratin between the nail plate and nail bed).
* Chronic plantar (moccasin) tinea pedis.
* History of current or past psoriasis of the skin and/or nails.
* Concurrent lichen planus.
* Onychogryphosis.
* Any of the following conditions of the great toenail:
* proximal subungual onychomycosis
* white superficial onychomycosis
* dermatophytoma or "yellow spike/streak"
* exclusively lateral disease
* confounding problems/abnormalities of the great toenail(s).
* Any abnormality that could prevent a normal appearing nail if clearing of infection is achieved.
* Inability for the toenail to become normal in the opinion of the investigator.
* History of multiple repeated failures with previous therapies for onychomycosis.
* Trauma to the affected great toenail(s).
* Use of oral antifungal agents in the past 6 months.
* Use of topical antifungal agents in the past 1 month.
* Prior surgical treatment of the affected great toe(s).
* Cancer and/or treatment of any type of cancer within the last six months.
* Peripheral vascular disease or peripheral circulatory impairment.
* History of uncontrolled diabetes mellitus.
* Known immunodeficiency.
* Known sensitivity, or contraindication, to light therapy.
* Pregnant, breast feeding, or planning pregnancy prior to the end of study participation.
* Serious mental health illness such as dementia or schizophrenia; psychiatric hospitalization in the past two years.
* Developmental disability or cognitive impairment that would preclude adequate comprehension of the informed consent form and/or ability to follow study subject requirements and/or record the necessary study measurements.
* Involvement in litigation and/or receiving disability benefits related in any way to the parameters of the study.
* Participation in a clinical study or other type of research in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Zang, DPM, Principal Investigator
Locations (1):
- Arizona Institute of Footcare Physicians, Mesa, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Erchonia FX-405™ Laser: The Erchonia FX-405™ Laser is a dual-diode laser emitting 15.5-17.5 milliWatts (mW) of 635 nanometer (nm) red laser light and 23.5-25.5 mW 405 nm blue laser light. The the power reaching the surface of the skin is 1 mW. The Erchonia FX-405™ Laser is activated such that the laser light is directed at the great toenail at a distance of approximately 6 inches above the toenail. The dual wavelengths of 405 nm and 635 nm are activated simultaneously for 10 minutes of total treatment administration time.
Period: Overall Study
Arm/Group | Erchonia FX-405™ Laser
Started | 105
Completed | 105
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia FX-405™ Laser
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (12.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 102
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 105
Percent (%) Toenail Onychomycosis Disease Involvement [Mean (Standard Deviation); unit: percent of toenail] — The percent (%) of the toenail that had onychomycosis disease involvement was determined.
  percent of toenail | 57.39 (21.86)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Toenails Attaining 25 Percent (%) or More Increase in Clear Nail
Description: Millimeter (mm) of clear nail from the base of the lunula was measured from digital photographs of the toenail using a computer program. Change in mm of clear nail bed was calculated as the difference in mm of clear nail bed from baseline measurement to the measurement at 3 months post-procedure administration. The percent (%) of increase in clear nail from baseline was calculated from there. An increase in mm or percent of clear nail between the two measurement points indicates the toenail onychomycosis has improved and is positive for study success. A decrease in mm or percent of clear nail between the two measurement points indicates the toenail onychomycosis has worsened and is negative for study success.
  Individual toenail success criteria was defined as 25 percent (%) or more increase in clear nail growth at 3 months post-procedure relative to baseline. Overall study success criteria was defined as 60% or more of treated toenails meeting the individual success criteria.
Time Frame: 12 weeks
Measure: Number; unit: percentage of toenails
Arm/Group | Erchonia FX-405™ Laser
Number analyzed (Participants) | 105
percentage of toenails | 65

2. Secondary Outcome: Change in Millimeter (mm) of Clear Nail Bed
Description: Millimeter (mm) of clear nail from the base of the toenail lunula was determined from digital photographs of the toenail using a computer program. Change in mm of clear nail bed was calculated as the difference in mm of clear nail bed from baseline measurement to the measurement at 3 months post-procedure administration. An increase in mm of clear nail between the two measurement points indicates that the toenail onychomycosis has improved and is positive for study success. A decrease in mm of clear nail between the two measurement points indicates that the toenail onychomycosis has worsened and is negative for study success.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: millilmeters
Arm/Group | Erchonia FX-405™ Laser
Number analyzed (Participants) | 105
millilmeters | 4.99 (2.24)
Statistical Analysis 1: Comparison: Erchonia FX-405™ Laser; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

3. Secondary Outcome: Change in Percent (%) of mm Clear Nail
Description: Millimeter (mm) of clear nail from the base of the lunula was measured from digital photographs of the toenail using a computer program. Change in mm of clear nail bed was calculated as the difference in mm of clear nail bed from baseline measurement to the measurement at 3 months post-procedure administration. The percent (%) of increase in clear nail from baseline was calculated from there.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of change in mm clear nail
Arm/Group | Erchonia FX-405™ Laser
Number analyzed (Participants) | 105
percentage of change in mm clear nail | 30.36 (19.43)
Statistical Analysis 1: Comparison: Erchonia FX-405™ Laser; results at 12 weeks compared to baseline; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Erchonia FX-405™ Laser
Serious Adverse Events (participants affected / at risk) | 0/105
Other Adverse Events (participants affected / at risk) | 0/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No